CLINICAL TRIAL: NCT02658487
Title: Phase II Trial of Vosaroxin in Combination With Infusional Cytarabine in Patients With Untreated AML
Brief Title: Vosaroxin and Infusional Cytarabine in Treating Patients With Untreated Acute Myeloid Leukemia
Acronym: VITAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sanjay Mohan, Assistant Professor of Medicine, Division of Hematology/Oncology, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC HEM 1553; NCI-2015-01735 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA068485 (NIH)
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Acute Myeloid Leukemia With Multilineage Dysplasia; Myeloid Sarcoma; Secondary Acute Myeloid Leukemia; Therapy-Related Acute Myeloid Leukemia; Therapy-Related Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Sarcoma, Myeloid | interventions — Cytarabine; vosaroxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (vosaroxin, cytarabine) (Experimental): Patients receive vosaroxin IV on days 1 and 4 and cytarabine IV continuously on days 1-7 (Induction I). Patients with residual leukemia and for whom a second course is indicated in the judgment of the investigator may undergo a second course of treatment (Induction II) 14-57 days after day 1 of Induction I.
  Interventions: Drug: Cytarabine; Drug: Vosaroxin

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Vosaroxin — Given IV
  Other Names: AG-7352; SNS-595; SPC 595; Voreloxin

SUMMARY:
This phase II trial studies how well vosaroxin and cytarabine work in treating patients with untreated acute myeloid leukemia. Drugs used in chemotherapy, such as vosaroxin and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the rate of complete remission (CR) after induction therapy with the combination of "7+V" (vosaroxin and standard dose infusional cytosine arabinoside [ara-C]) for patients with newly diagnosed, previously untreated acute myelogenous leukemia (AML).

SECONDARY OBJECTIVES:

I. Frequency of grade 3-5 adverse events related to administration of "7+V".

II. To evaluate for the presence of minimal residual disease (MRD) remaining after "7+V" induction and/or re-induction.

III. To determine the CR/CR with incomplete blood count recovery (CRi) rate after one and/or 2 cycles of "7+V" induction.

IV. To determine the time to neutrophil and platelet recovery following "7+V" induction.

V. To assess disease-free survival (DFS) at 1 year (yr) of patients achieving CR/CRi after "7+V" induction.

VI. To assess overall survival (OS) at 1 yr of all patients receiving protocol-defined therapy.

VII. To determine the correlation of hematopoietic stem cell transplant (HSCT) comorbidity index and Wheatley Index scores with disease response, DFS and OS.

TERTIARY OBJECTIVES:

* I. To describe the mutational burden of this cohort of AML patients.
* II. To correlate genomic aberration with response rate, DFS, and OS.
* III. To determine the number of patients treated with vosaroxin who eventually go to allogeneic HSCT.

OUTLINE:

Patients receive vosaroxin intravenously (IV) on days 1 and 4 and cytarabine IV continuously on days 1-7 (Induction-I). Patients with residual leukemia and for whom a second course is indicated in the judgment of the investigator may undergo a second course of treatment (Induction-II) 14-57 days after day 1 of Induction-1

After completion of study treatment, patients are followed every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Ability to tolerate intensive therapy with vosaroxin 90 mg/m^2 and cytarabine
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 at time of study entry
* Morphologically confirmed new diagnosis of AML in accordance with World Health Organization (WHO) diagnostic criteria
* Patients who have received hydroxyurea alone or have previously received "non-cytotoxic" therapies for myelodysplastic syndromes (MDS) or myeloproliferative neoplasms (MPN) (e.g., thalidomide or lenalidomide, 5-azacytidine or decitabine, histone deacetylase inhibitors, low-dose Cytoxan, tyrosine kinase or dual tyrosine kinase [TK]/SRC proto-oncogene, non-receptor tyrosine kinase [src] inhibitors) will be allowed
* Serum creatinine =< 2.0 mg/dL
* Hepatic enzymes (alanine aminotransferase [ALT], aspartate aminotransferase [AST]) =< 2.5 x upper limit of normal
* Total bilirubin =< 1.5 x upper limit of normal unless clearly related to Gilbert's disease, hemolysis or leukemic infiltrate
* FOR PATIENTS IN STAGE 1 (PATIENTS #1-#17)
* >= 55 years of age with AML of any risk classification, or 18-54 years of age with high-risk AML disease based on one of the following:

  * Antecedent hematologic disorder including myelodysplasia (MDS)-related AML (MDS/AML) and prior myeloproliferative disorder (MPD)
  * Treatment-related myeloid neoplasms (t-AML/t-MDS)
  * AML with FMS-like tyrosine kinase 3 (FLT3) - internal tandem duplication (ITD)
  * Myeloid sarcoma
  * AML with multilineage dysplasia (AML-MLD)
  * Adverse cytogenetics (defined as -5/-5q; -7/-7q; abnormal 3q, 9q, 11q, 20q, 21q or 17p; t(6;9); t(9;22); trisomy 8; trisomy 13; trisomy 21; complex karyotypes (>= 3 clonal abnormalities); monosomal karyotypes
* FOR PATIENTS IN STAGE 2 (ENROLLED PATIENT #18 AND BEYOND)
* >= 55 years of age with AML of any risk classification, or 18-54 years of age with intermediate or high risk AML as defined by National Comprehensive Cancer Network (NCCN) risk assignment

Exclusion Criteria:

* STAGES 1 AND 2
* Patients with acute promyelocytic leukemia (APL) as diagnosed by morphologic criteria, flow cytometric characteristics, and rapid cytogenetics or fluorescence in situ hybridization (FISH) or molecular testing
* Any previous treatment with vosaroxin
* Concomitant chemotherapy, radiation therapy

  * For patients with hyperleukocytosis with > 50,000 blasts/μL; leukapheresis or hydroxyurea may be used prior to study drug administration for cytoreduction at the discretion of the treating physician
* Active, uncontrolled infection

  * Patients with infection under active treatment and controlled with antibiotics, antivirals, or antifungals are eligible
  * Chronic hepatitis is acceptable
* Active, uncontrolled graft vs. host disease (GVHD) following allogeneic transplant for non-AML condition (e.g. MDS, lymphoid malignancy, aplastic anemia); patients with GVHD controlled on stable doses of immunosuppressants are eligible
* Presence of other life-threatening illness
* Left ventricular ejection fraction (LVEF) < 40% as measured by echocardiogram or multi gated acquisition scan (MUGA)
* Known or suspected central nervous system (CNS) involvement of active AML
* Other active malignancies including other hematologic malignancies or other malignancies within 12 months before randomization, except nonmelanoma skin cancer or cervical intraepithelial neoplasia
* History of myocardial infarction (MI), unstable angina, cerebrovascular accident, or transient ischemic attack (CVA/TIA) within 3 months before randomization
* Prior or current therapy:

  * Hydroxyurea or medications to reduce blast count within 24 hours before randomization
  * Treatment with an investigational product within 14 days before randomization, or not recovered from all acute effects of previously administered investigational products
* Renal insufficiency requiring hemodialysis or peritoneal dialysis
* Pregnant or breastfeeding
* Known human immunodeficiency virus (HIV) seropositivity
* Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the investigator or medical monitor
* ADDITIONAL EXCLUSION CRITERIA APPLIED TO STAGE 1
* Patients 18-54 years of age with "good risk" AML defined as the presence of t(8;21), inv(16), or t(16;16) as diagnosed by morphologic criteria, flow cytometric characteristics, and rapid cytogenetics or FISH
* Patients with t(8;21), inv(16), t(16;16) who are unable to receive anthracycline based induction will be allowed to enroll provided the medical reason they are unable to receive anthracyclines is clearly documented and provided they fulfill all other eligibility and criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-03; Primary Completion 2019-04 (Actual); Study Completion 2024-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Mohan, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center; Michael Savona, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - Medical University of South Carolina Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this trial was March 2016 to April 2019. Participants were recruited at Vanderbilt University Medical Center, Yale University, and University Medical School, South Carolina.
Pre-assignment Details: 42 participants met all eligibility criteria and were enrolled on this study. Nine of the participants received a second induction.
Groups:
- Treatment (Vosaroxin, Cytarabine) Induction: Patients receive vosaroxin IV on days 1 and 4 and cytarabine IV continuously on days 1-7 (Induction I). Patients with residual leukemia and for whom a second course is indicated in the judgment of the investigator may undergo a second course of treatment (Induction II) 14-57 days after day 1 of Induction I.
  Cytarabine: Given IV
  Vosaroxin: Given IV
Period: Overall Study
Arm/Group | Treatment (Vosaroxin, Cytarabine) Induction
Started | 42
Completed | 26
Not Completed | 16
Not completed — Death | 2
Not completed — Disease progression | 10
Not completed — Alternative therapy | 1
Not completed — Adverse Event | 1
Not completed — Treatment Failure, circulating blasts | 1
Not completed — Refractory acute myeloid leukemia (AML) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Vosaroxin, Cytarabine)
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 17
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 64.4 [33.4 to 74.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35
  Black or African American | 5
  Unknown/unreported | 2
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate (CR)
Description: CR is calculated as the percentage of patients with complete remission after the therapy. The response criteria is based on International Working Group Criteria. Complete Remission: Neutrophils(cells/μl)>1000, Platelets (plt/μl)≥ 100,000,Bone marrow blasts (%) <5; CR with incomplete count recovery (CRi): meets criteria for CR except for neutrophils ≤1000 or Meets criteria for CR except for platelets< 100,000; Partial Remission: CR except for Bone marrow blasts (%) Decrease of ≥ 50% to value between 5% and 25%; Treatment Failure:Persistent acute myeloid leukemia in blood or bone marrow, or therapy fails to achieve a remission of any category, or death prior to response assessment
Time Frame: Up to 3 months
Population: Evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Vosaroxin, Cytarabine)
Number analyzed (Participants) | 42
Participants | 20

2. Secondary Outcome: Event-free Survival
Description: Survival distribution will be estimated using the method of Kaplan and Meier. Event-free survival time is defined as the time from start of therapy to progression or death for any reason (which ever comes first), and those alive without progression are censored at the last day of follow up.
Time Frame: From start of therapy up to 1 year
Population: All patients participated
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Vosaroxin, Cytarabine)
Number analyzed (Participants) | 42
months | 7.6 [2.9 to NA] — insufficient number of participants with events for estimating

3. Secondary Outcome: Frequency of Grade 3-5 Adverse Event Related to Cytarabine and Vosaroxin (7+V)
Description: Events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Counts of all events are summed up.
Time Frame: Up to 3 months
Population: All participants
Measure: Number; unit: adverse events
Arm/Group | Treatment (Vosaroxin, Cytarabine)
Number analyzed (Participants) | 42
adverse events | 133

4. Secondary Outcome: Leukemia-free Survival (LFS or DFS)
Description: Survival distribution will be estimated using the method of Kaplan and Meier. LFS time is defined as the time from complete remission to disease progression or death for any reason and those disease free and alive are censored at the last day of follow up.
Time Frame: The time from complete remission to disease progression or death for any reason, assessed up to 1 year
Population: Patients who had complete remission after the therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Vosaroxin, Cytarabine)
Number analyzed (Participants) | 20
months | NA [13.1 to NA] — the median and upper bound are not estimable due to not long enough follow up

5. Secondary Outcome: Overall Survival
Description: Survival distribution will be estimated using the method of Kaplan and Meier. The overall survival time is defined as time from start of therapy to death of any reason. Those alive are censored at the last day of known alive.
Time Frame: The time from start of therapy to death, assessed up to 1 year
Population: All participated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Vosaroxin, Cytarabine)
Number analyzed (Participants) | 42
months | 10.7 [7.4 to NA] — insufficient number of participants with events for estimating the upper bound

6. Secondary Outcome: Minimal Residual Disease
Description: Frequency of minimal residual disease (MRD) remaining after "7+V" induction and/or re-induction
Time Frame: Up to 3 months
Population: When this study was designed, it was anticipated that the data needed to calculate MRD was going to be available from standard of care. However, this ended up not being the case. MRD requires NGS testing and the study did not have budget to cover this testing. Since the NGS was not part of the standard of care for these patients, these data were not available to collect as part of the study. There is no intention to go back and report data for this Outcome Measure if funding became available.
Arm/Group | Treatment (Vosaroxin, Cytarabine) Induction
Number analyzed (Participants) | 0

7. Secondary Outcome: Rate of CR/CRi
Description: Frequency of Complete Remission / Complete Remission with Incomplete Count Recovery (CR/CRi) after "7+V" induction and/or re-induction
Time Frame: Up to 3 months
Population: Evaluable patients
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Treatment (Vosaroxin, Cytarabine)
Number analyzed (Participants) | 42
Proportion of participants | 0.55 [0.40 to 0.69]

8. Other Pre Specified Outcome: Correlation of Three Standard Prognostic Scores of AML Risk With Disease Response
Description: Correlate hematopoietic stem cell transplant (HSCT) comorbidity index, Wheatley Index, and AML-Score values with disease response
Time Frame: Up to 3 months
Population: Data for this outcome measure were not collected.
Arm/Group | Treatment (Vosaroxin, Cytarabine)
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Correlate HSCT Comorbidity Index, Wheatley Index, and AML-Score Values With DFS
Description: Correlation of three standard prognostic scores of AML risk with disease free survival
Time Frame: The time from complete remission to disease progression or death for any reason, assessed up to 1 year
Population: Data for this outcome measure were not collected.
Arm/Group | Treatment (Vosaroxin, Cytarabine)
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Correlation of Standard Prognostic Scores of AML Risk With Survival
Description: Correlate HSCT comorbidity index, Wheatley Index, and AML-Score values with overall survival
Time Frame: The time from start of therapy to death for any reason, assessed up to 1 year
Population: Data for this outcome measure were not collected.
Arm/Group | Treatment (Vosaroxin, Cytarabine)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events that emerge (or worsen) after the first dose of study drug and within 30 days after the last dose.
Groups:
- Treatment (Vosaroxin, Cytarabine) Induction 1: Patients receive vosaroxin IV on days 1 and 4 and cytarabine IV continuously on days 1-7 (Induction I).
  Cytarabine: Given IV
  Vosaroxin: Given IV
- Induction 2: Patients with residual leukemia and for whom a second course is indicated in the judgment of the investigator may undergo a second course of treatment (Induction II) 14-57 days after day 1 of Induction I.
Arm/Group | Treatment (Vosaroxin, Cytarabine) Induction 1 | Induction 2
All-Cause Mortality (participants affected / at risk) | 18/33 | 4/9
Serious Adverse Events (participants affected / at risk) | 10/33 | 5/9
Other Adverse Events (participants affected / at risk) | 33/33 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vosaroxin, Cytarabine) Induction 1 (N=33) | Induction 2 (N=9)
Altered mental state (Psychiatric disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Acute sigmoid diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 3 (4) | 0 (0)
Colitis (Gastrointestinal disorders) | 6 (8) | 1 (1)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Fungemia (Infections and infestations) | 1 (1) | 0 (0)
Chronic heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Thromboembolic event - Related to Hickman line placement (Vascular disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vosaroxin, Cytarabine) Induction 1 (N=33) | Induction 2 (N=9)
Anemia (Blood and lymphatic system disorders) | 10 (10) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 27 (33) | 5 (10)
Creatinine increased (Investigations) | 2 (6) | 0 (0)
Neutrophil count decreased (Investigations) | 17 (36) | 4 (8)
Platelet count decreased (Investigations) | 21 (55) | 5 (20)
Urine output decreased (Investigations) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 16 (29) | 5 (16)
Colitis (Gastrointestinal disorders) | 5 (5) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 26 (37) | 5 (19)
Mucositis oral (Gastrointestinal disorders) | 11 (20) | 5 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5) | 2 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Confusion (Psychiatric disorders) | 3 (3) | 0 (0)
Bacteremia/multiorgan failure (Infections and infestations) | 0 (0) | 1 (1)
Catheter related thorombosis (Vascular disorders) | 0 (0) | 1 (1)
Concern for fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic colitis (Investigations) | 0 (0) | 1 (1)
Staph bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 (4)
Transaminitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Worsening Platelet Count Decrease (Investigations) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Soft Tissue Infection (Infections and infestations) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT02658487/Prot_SAP_000.pdf